CLINICAL TRIAL: NCT04014335
Title: An Open-Label Phase 2a Clinical Study to Evaluate the Effectiveness and Safety of IONIS-FB-LRx, an Antisense Inhibitor of Complement Factor B, in Adult Subjects With Primary IgA Nephropathy
Brief Title: A Study to Evaluate the Effectiveness and Safety of IONIS-FB-LRx, an Antisense Inhibitor of Complement Factor B, in Adult Participants With Primary IgA Nephropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISIS 696844-CS4
Record Dates: First submitted 2019-07-08; First posted 2019-07-10 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Primary IgA Nephropathy
MeSH Terms: conditions — Glomerulonephritis, IGA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- IONIS-FB-LRx (Experimental)
  Interventions: Drug: IONIS-FB-LRx

INTERVENTIONS:
Drug: IONIS-FB-LRx — Participants will receive IONIS-FB-LRx, by subcutaneous injection (SC) at Week 1 and every 4 weeks through Week 25. Optional 48-week Extension, with drug dosing continuing every 4 weeks.

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of IONIS-FB-LRx, an antisense inhibitor of complement factor B messenger ribonucleic acid (CFB mRNA), and to evaluate the effect of IONIS-FB-LRx on plasma factor B (FB) levels and serum AH50, CH50 activity in participants with primary immunoglobulin A (IgA) nephropathy.

DETAILED DESCRIPTION:
This is a Phase 2, single arm open-label clinical study in up to 25 participants that will consist of a screening period, a 24-week treatment period, an optional treatment extension period of up to an additional 48 weeks, and a 12- week post-treatment follow-up evaluation period.

ELIGIBILITY:
Inclusion Criteria

* Females must be non-pregnant and non-lactating, and either surgically sterile or post-menopausal OR use a highly effective method of birth control
* Biopsy-proven primary immunoglobulin A (IgA) nephropathy
* Hematuria
* Proteinuria

Exclusion Criteria

* Clinically significant abnormalities in medical history (e.g., dementia, stroke, acute coronary syndrome, thrombocytopenia, or major surgery within 3 months of Screening)
* Diagnosis of primary or secondary immunodeficiencies of B-lymphocyte function, splenectomy, or history of recurrent meningococcal disease
* Active infection 30 days prior to study
* Estimated glomerular filtration rate (eGFR) ≤ 40 milliliters per minute per 1.73 square meters (mL/min/1.73m^2) using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI)
* Presence of another renal disease including, but not limited to, diabetes and/or diabetic nephropathy, thin basement membrane disease, Alport's disease, IgA Nephritis (Henoch-Schonlein purpura), lupus nephritis, Minimal Change Disease, post-infectious glomerulonephritis or any other cause of proteinuria or secondary IgA nephropathy (including, but not limited to Celiac disease, Crohn's disease, human immunodeficiency virus (HIV), liver cirrhosis)
* History of renal transplant or another organ transplant
* Treatment with another investigational drug, biological agent, or device within 6 months of screening, or 5 half-lives of investigational agent, whichever is longer
* Administration of immunosuppressive/immunomodulatory medication 12 months prior to study drug administration, except for short-term treatments.
* Other protocol-specified inclusion/exclusion criteria may apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2019-12-04 (Actual); Primary Completion 2024-02-08 (Actual); Study Completion 2024-04-11 (Actual)

PRIMARY OUTCOMES:
Percent Reduction in 24-hour Urine Protein Excretion | Baseline to Week 29 (If participant discontinues Study Drug prior to Week 25, Baseline and 4 weeks after the last dose of Study Drug will be measured)

SECONDARY OUTCOMES:
Absolute Reduction in 24-hour Urine Protein Excretion | Baseline to Week 29 (If participant discontinues Study Drug prior to Week 25, Baseline and 4 weeks after the last dose of Study Drug will be measured)
Absolute Reduction in Albuminuria (UACr Ratio) | Baseline to Week 29
Absolute Reduction in Proteinuria (UPCr Ratio) | Baseline to Week 29
Percent Change from Baseline in Plasma Factor B (FB) | Up to Week 29
Percent Change from Baseline in Plasma AH50 | Up to Week 29

CONTACTS AND LOCATIONS:
Locations (7):
- Australia (3):
  - IONIS Investigative Site, Liverpool, New South Wales
  - IONIS Investigative Site, St Leonards, New South Wales
  - IONIS Investigative Site, Parkville, Victoria
- Canada (2):
  - IONIS Investigative Site, Vancouver, British Columbia
  - IONIS Investigative Site, Toronto, Ontario
- IONIS Investigative Site, Christchurch, New Zealand
- IONIS Investigative Site, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Barbour SJ, Hladunewich MA, McCaleb ML, Robson R, Barrett TD, Yin L, Frazer-Abel A, Garg JP, Geary R, Schneider E, Brice GT. A single-arm phase 2 trial of an investigational RNA therapeutic to complement factor B sefaxersen for treatment of IgA nephropathy. Kidney Int. 2025 Dec 22:S0085-2538(25)01007-5. doi: 10.1016/j.kint.2025.11.017. Online ahead of print. PMID 41443406
- [Derived] Tekendo-Ngongang C, Gleeson JG, Mignon L. Treating the Untreatable: Antisense Oligonucleotides as an Individualized Therapy for Rare Genetic Kidney Diseases. J Am Soc Nephrol. 2024 Dec 1;35(12):1774-1777. doi: 10.1681/ASN.0000000532. Epub 2024 Sep 27. No abstract available. PMID 39331470